CLINICAL TRIAL: NCT03612349
Title: Assessing Tobacco Product Choice When the Cost of Menthol Cigarettes Increases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1708001884
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Tobacco Use; Cigarette Smoking
Keywords: cigarettes; smoking
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking; Smoking

STUDY DESIGN:
Intervention Model Description: Participants will complete the Experimental Tobacco Marketplace Task under two marketplace conditions. One condition has all tobacco products available in menthol and non-menthol flavors. The other condition does not include alternative flavored combusted products.
Masking Description: There is no masking since participants experience both marketplace conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Condition 1: All Products (Other): Experimental Tobacco Marketplace Task is a behavioral economics task. During the task, participants purchase products from an online tobacco marketplace. In this condition, all tobacco products are available in menthol and non-menthol flavors.
  Interventions: Behavioral: Experimental Tobacco Marketplace Task
- Condition 2: No menthol LCCs (Other): Experimental Tobacco Marketplace Task is a behavioral economics task. During the task, participants purchase products from an online tobacco marketplace. In this condition, the online tobacco marketplace does not include menthol flavored little cigars and cigarillos.
  Interventions: Behavioral: Experimental Tobacco Marketplace Task

INTERVENTIONS:
Behavioral: Experimental Tobacco Marketplace Task — Participants will select tobacco products from an Experimental Online Tobacco Marketplace under both marketplace conditions.
  Other Names: Condition 1: All Products; Condition 2: No menthol LCCs

SUMMARY:
In this study, participants will complete a behavioral economics laboratory task and validation field assessments to understand how menthol cigarette policy restrictions may affect tobacco product purchasing and use.

DETAILED DESCRIPTION:
We will enroll 60 smokers who will complete four lab sessions and two field assessments. Participants meeting initial eligibility criteria over the phone will complete an in-person screening visit. Breath carbon monoxide and alcohol tests will be collected. Participants will answer questionnaires on the computer and via interview about their tobacco use and medical history. Eligible participants will remain in the lab to complete additional baseline questionnaires and will be given the opportunity to sample alternative tobacco products, such as LCCs, smokeless tobacco, electronic cigarettes, and nicotine replacement.

During the next two lab sessions, participants will complete a behavioral economics assessment, the Experimental Tobacco Marketplace task, designed to simulate purchasing tobacco products online. Participants will be given 'coupons' to obtain tobacco products from the online experimental marketplace. After these lab sessions, participants will be provided with the tobacco products they selected from the online experimental marketplace to use during 3-day field assessments to validate the task. Participants will be told to only use tobacco products provided by the lab during the field assessments. At both lab sessions, participants will complete questionnaires about their tobacco use, mood, and reactions to the alternative tobacco products. At the final lab session, a qualitative interview will be conducted to learn more about the participants' experiences selecting and using tobacco products.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 and older
2. Daily smokers who smoke on average at least 5 cigarettes per day for the past 12 months
3. Self-report smoking a menthol cigarette brand
4. Must report use of an alternative tobacco product(s) at least once in the past month
5. Breath CO levels > 8 ppm (if < 8 ppm, then NicAlert Strip = 6)
6. Speak, comprehend, and read English well enough to complete study procedures

Exclusion Criteria:

1. Breath alcohol level > 0.01 ng/ml
2. Intention to quit smoking in the next 30 days
3. Self-reported serious medical or psychiatric conditions during the past 12 months including:

   1. heart attack
   2. stroke
   3. angina
   4. blood clots in the arms or legs for which the individual is undergoing active medical treatment
   5. cancer requiring active chemotherapy or radiation therapy
   6. chronic obstructive pulmonary disease
   7. schizophrenia
4. Pregnant or breastfeeding
5. CO reading > 80 ppm
6. Enrollment stratum (white or African-American/black) is full

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Total amount of combusted tobacco purchased in mg of nicotine. | through study completion, an average of 2-weeks.
  How much combusted tobacco is purchased by the participants.

SECONDARY OUTCOMES:
Tobacco Product Demand Curves | through study completion, an average of 2-weeks.
  Purchasing data will be used to generate demand curves for each tobacco product available on the online tobacco marketplace.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Denlinger, MPH, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No